CLINICAL TRIAL: NCT00382759
Title: Nonmyeloablative Allogeneic Stem Cell Transplantation in Elderly Patients With Hematological Malignancies:Results From the GITMO (Gruppo Italiano Trapianto Midollo Osseo)Multicenter Prospective Clinical Trial
Brief Title: Nonmyeloablative Stem Cell Transplant in Elderly
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012000
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: stem cell transplant

SUMMARY:
The study aimed to evaluate the efficacy of a nonmyeloablative conditioning consisting of fludarabine and total body irradiation in patients older than 60 years of age

DETAILED DESCRIPTION:
A total of 35 patients with hematological malignancies were treated with fludarabine (30 mg/m2 x 3-5 days) and 200 cCy TBI followed by allogeneic hematopoietic stem cell transplantation (HSCT) from a matched-sibling donor.

Neutrophil recovery occurred in 89% of the patients at a median time of 15 days. On day +30, 10 patients had > 95% donor chimerism, and 21 patients had mixed chimerism. The cumulative probabilities of grade II-IV acute GVHD and chronic GVHD were 51% and 84% respectively. Transplant-related mortality at 100 days and 1 year was 5% and 9% respectively. The probabilities of 1-year overall (OS) and progression-free survival (PFS) were 55% and 47% respectively. The estimated 1-year probability of OS and PFS for patients in early disease stages were 87% and 74% respectively , which were significantly higher than the survival and PFS estimates of 12% obtained in patients with advanced disease stages at the time of transplant

ELIGIBILITY:
Inclusion Criteria:

* patients with myeloid or lymphoid malignancy who were > 60 years old potentially treatable with stem cell transplant

Exclusion Criteria:

* lack of an HLA-identical sibling donor

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2000-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
overall survival
progression-free survival
transplant-related mortality

SECONDARY OUTCOMES:
acute GVHD
chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: michele falda, md, Principal Investigator — ospedale san giovanni battista
Locations (1):
- Ospedale San Giovanni Battista, Torino, Italy